CLINICAL TRIAL: NCT04321213
Title: In-hospital Healthcare Professionals' Attitudes and Their Experience in Performing Cardiopulmonary Resuscitation.
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Region Västmanland (Other); Dalarna University (Other); Center for Clinical Research Dalarna, Sweden (Other)
Responsible Party: Principal Investigator, Jennie Silverplats, Principal investigator, Dalarna County Council, Sweden
Other Study IDs: 2006/201/2 (part 2)
Record Dates: First submitted 2020-02-21; First posted 2020-03-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: In-hospital Cardiac Arrest
Keywords: in-hospital cardiac arrest; attitudes; cardiopulmonary resuscitation; CPR
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare professionals in the Region of Västmanland: Healthcare professionals of all professions working in-hospital with patient contact at two hospitals in the Region of Västmanland, Sweden. Data is collected by questionnaires.
- Healthcare professionals in the Region of Dalarna: Healthcare professionals of all professions working in-hospital with patient contact at three hospitals in the Region of Dalarna, Sweden. Data is collected by questionnaires.

SUMMARY:
Attitudes among healthcare professionals can possibly affect the treatment given in cardiac arrest situations. The attitudes of healthcare professionals towards cardiopulmonary resuscitation (CPR) has been poorly studied. The few existing previous international results shows attitudes reported by nurses as hesitation, fear of defibrillation, anxiety and fear of harming the patient.

The aim of this study was to describe the attitudes towards performing cardiopulmonary resuscitation among in-hospital healthcare professionals, furthermore to assess if experience in performing CPR has an effect on attitudes.

DETAILED DESCRIPTION:
Data will be collected using questionnaires containing attitude questions. The questionnaires contains questions regarding attitudes towards being required to perform CPR (6 questions), previous experience in performing CPR (time since last performance and number of performances) and attitudes during the latest CPR performance (8 questions). All attitude questions are constructed as multiple choice questions.

Results regarding attitudes towards being required to perform CPR and attitudes during the latest CPR performance will be presented descriptively. To analyse a possible effect of time since CPR performance and number of CPR performances on attitudes during the latest CPR performance logistic regression will be used. Response variables will be "yes" or "no" on 8 specific attitude questions with predictors consisting of time since CPR performance (0-3 months ago, 4-23 months ago and >24 months) and number of CPR performances (1-3 times, 4-10 times and >10 times).

ELIGIBILITY:
Inclusion Criteria:

* In-hospital healthcare professionals.
* Patient contact

Exclusion Criteria:

* Absent during the survey
* Parental leave
* Leave of absence
* Sick leave.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital healthcare professionals of all professions at five hospitals in the region of Västmanland and Region of Dalarna, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 3639 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
In-hospital healthcare professionals' attitudes towards CPR. | one month
  14 questions regarding attitudes towards performing CPR will be presented descriptively. Number of respondents answering "yes", "no" and "I don´t know" to each attitude question will be presented.
In-hospital healthcare professionals' experience in performing CPR. | one month
  Two questions regarding experience in performing CPR will be presented descriptively. Number of respondents in each response category concerning number of previous CPR performances and time since last CPR performance will be presented.
Does experience in performing CPR have an effect on attitudes towards CPR | two months
  The effect of previous experience in CPR on attitudes during a cardiac arrest situation will be analysed using binary logistic regression. Each of the eight questions concerning attitudes during a cardiac arrest situation will serve as a dependent variable with "yes" as the response. Independent variables consists of number of previous CPR performances, time since last CPR performance and workplace. Independent variables associated with the dependent variable at a level of p <0.1 will be included in a multiple model. The model will be adjusted for profession and number of years in profession.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Strömsöe, PhD, Study Director — Dalarna County Council
Locations (2):
- Sweden (2):
  - Region of Västmanland, Västerås, Västmanland County
  - Region of Dalarna, Mora

IPD SHARING:
Plan to Share IPD: No